CLINICAL TRIAL: NCT03815721
Title: Carry-over Effects of Repetitively Applied Transcutaneous Spinal Cord Stimulation on Spasticity and Residual Motor Control in Incomplete Spinal Cord Injured Individuals
Brief Title: Carry-over Effects of Repetitively Applied Transcutaneous Spinal Cord Stimulation on Spasticity
Acronym: SCS-CorE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study terminated by the PIs due to unexpected outcomes
Sponsor: Swiss Paraplegic Research, Nottwil (Network)
Collaborators: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Bersch-Porada Ines, PhD in Medical Sciences, Swiss Paraplegic Research, Nottwil
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2016-16
Record Dates: First submitted 2019-01-22; First posted 2019-01-24 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Spinal Cord Injuries; Spasticity, Muscle
MeSH Terms: conditions — Spinal Cord Injuries; Muscle Spasticity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- daily stimulation (Experimental): 30-minute sessions of transcutaneous spinal cord stimulation using the Stimulette r2x+ will be repetitively applied 7 times per week.
  Interventions: Device: Stimulette r2x+
- stimulation every other day (Experimental): 30-minute sessions of transcutaneous spinal cord stimulation using the Stimulette r2x+ will be repetitively applied 3 times per week.
  Interventions: Device: Stimulette r2x+

INTERVENTIONS:
Device: Stimulette r2x+ — device for repetitive transcutaneous spinal cord stimulation

SUMMARY:
Spinal cord injury is a devastating condition, causing substantial impairment of vital body functions caudal to the lesion. A major cause of disability stems from spasticity, a common secondary sequelae. Its various clinical manifestations include spasms, clonus, and resistance to passive movements, and often present a major hindrance in rehabilitation, further deteriorate residual motor performance, and negatively impact independence and quality of life. Despite its high prevalence, successful management of spasticity has remained difficult. Standard-of-care treatment modalities are often insufficient or bear the risk of undesirable side effects further accentuating paresis. Epidural stimulation of the lumbar spinal cord via implanted electrodes provides for an alternative approach. It works through modifying the dysregulated neural signal processing of spared spinal circuitry caudal to the injury. Its ameliorative effects on severe lower-limb spasticity have been repetitively reported. Yet, epidural spinal cord stimulation in motor disorders is still off-label, applied in relatively few patients only, also because of its invasive character, the time consuming testing phase for its effective application, and the lack of markers to identify responders in advance. With the development of transcutaneous spinal cord stimulation, a method became available to activate the same input structures to the lumbar spinal cord as with epidural stimulation and hence to induce similar neuromodulatory effects, yet non-invasively, using standard equipment available at rehabilitation centers. A recent proof-of-concept study has shown that a single 30-minute session of transcutaneous spinal cord stimulation controlled various clinical signs of spasticity and augmented residual motor control in spinal cord injured individuals for several hours beyond its application. Further, in one subject, the stimulation was repetitively applied for six weeks, resulting in cumulative therapeutic effects persisting for 10 days after its discontinuation. These observations strongly suggest that the stimulation can induce beneficial neuroplastic adaptations of spared spinal systems and their interaction with residual supraspinal control. The proposed research aims at studying the reproducibility of these findings in a statistically sound cohort of individuals with spinal cord injury and testing the applicability and acceptance of transcutaneous spinal cord stimulation as a home-based therapy.

ELIGIBILITY:
Inclusion Criteria:

* motor and sensory incomplete spinal cord injury classified as grade C or D on the American Spinal Injury Association Impairment Scale
* neurological level of spinal cord injury: third cervical to tenth thoracic segment
* chronic condition (≥ 12 months post-spinal cord injury)
* preserved segmental and cutaneo-muscular reflexes in the lower limbs
* able to be verticalized for 6 minutes (with walking aids)
* preserved joint mobility, no musculoskeletal diseases
* spasticity (with/without antispasticity medication)
* stable antispasmodic medication one month prior to as well as during study participation

Exclusion Criteria:

* neuromuscular diseases, e.g., amyotrophic lateral sclerosis (ALS), Parkinson's disease, Guillain-Barré syndrome, muscular dystrophy
* dermatological issues at the stimulation site
* acute urinary tract infection at study entry
* active implants (e.g., cardiac pacemaker, drug pump)
* passive implants between the ninth thoracic level and the first lumbal level (e.g. metal screws/plates for surgical stabilization of spinal fractures)
* malignant diseases
* heart insufficiency
* potential pregnancy (pregnancy test to be conducted as part of the first evaluation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2021-05-10 (Actual); Study Completion 2021-05-10 (Actual)

PRIMARY OUTCOMES:
Change in spasticity index | from day 1 to day 57
  Spasticity index based on the Wartenberg pendulum test: For the pendulum test, subjects will be in a supported sitting position with the trunk reclined approximately 30°. The examiner will lift one leg to a horizontal position, release it, and let it oscillate passively until it stops. The pendulum test will be repeated three times on each side, separated by phases of relaxation. The spasticity index is calculated subtracting the knee angle of the initial horizontal leg position from the peak flexion angle of the first swing divided by the final knee resting angle. Scores ≥ 1 denote non-spastic conditions, and 0 extreme spasticity.

SECONDARY OUTCOMES:
Change in numeric rating scale spasticity | day 1, 8, 29, 50 and 57
  The severity of spasticity is rated using a numeric rating scale from a minimum of 0 to a maximum of 10. Higher values represent worse outcome.
Change in Modified Ashworth Scale | from day 1 to day 57
  The resistance to passive movement will be clinically graded according to the Modified Ashworth Scale. Individual scores from both legs will be summed (with a value of 1.5 for the 1+ scoring category) to result in a single Modified Ashworth Scale-sum score (0-96; 0, no increase in muscle tone) per assessment. Higher values represent worse outcome.
Change in adductor tone rating | from day 1 to day 57
  5-point ordinal scale describing adductor tone during passive abduction (0: normal tone - 4: maximal tone). Higher values represent worse outcome.
Change in Penn Spasm Frequency Scale | from day 1 to day 57
  5-point scale rating the frequency and severity of spasms (0: no spasms - 4: more than 10 spasms per hour). Higher values represent worse outcome.
Change in resistance of the lower limbs | from day 1 to day 57
  Measure of the resistance of the lower limbs to manipulation performed by a robotic system (MotionMaker, SWORTEC SA). The MotionMaker measures torque (N) and power output (W).
Change in 6-minute walk test | from day 1 to day 57
  distance in meters walked over a span of 6 minutes
Change in Walking Index for Spinal Cord Injury II Scale | from day 1 to day 57
  21-point ordinal scale that rates the extent and nature of assistance (e.g., walker, crutches, cane, braces, physical assistance) required to complete the 10-m walk test (0: unable to complete the test - 20: ambulated without any assistance). Higher values represent better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Ursula Hofstötter, Principal Investigator — Medical University Vienna; Angela Frotzler, Principal Investigator — Swiss Paraplegic Centre
Locations (1):
- Swiss Paraplegic Centre, Nottwil, Canton of Lucerne, Switzerland

IPD SHARING:
Plan to Share IPD: No